CLINICAL TRIAL: NCT04138108
Title: The Effect of Psychoeducation on Stress in Parents of Children With Attention Deficit Hyperactivity Disorder (ADHD): A Randomized Controlled Study
Brief Title: Psychoeducation in Parents of Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Gül Dikec, Assistant Professor in Nursing, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GO2017/9
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: ADHD; Parents
Keywords: Childhood illness; Stress; Parents; Psychiatric Nursing
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Two sessions of psychoeducation were given to the parents in the experimental group.
  Interventions: Other: Psychoeducation
- Control Group (No Intervention): The parents in the control group did not undergo any intervention and the children of the parents in this group continued their current treatment plans.

INTERVENTIONS:
Other: Psychoeducation — The parents of each child were educated as couples and each training session lasted 45-60 minutes for each family. Approximately the first five minutes of the training were used for warm-up, 25 minutes were used for basic ADHD knowledge and the last 15 minutes were catechetic and conducted interactively. The psychoeducation included discussion about the causes, symptoms and signs of ADHD, the course and characteristics of the disease according to age, the treatment process, the drugs used in the treatment and their side effects, correct and incorrect information about drugs, the other symptoms which can coexist with ADHD and their treatment, and what the parents can do about these issues.
  Arms: Experimental Group

SUMMARY:
The objective of this study was to determine the effect of psychoeducation on the stress levels of parents of children with Attention Deficit and Hyperactivity Disorder (ADHD). This was a randomised controlled study and applied the Consolidated Standards of Reporting Trials (CONSORT) statement. A total of 172 parents (experimental group: 86, control group: 86) participated in the study, which was planned as an experimental (randomized controlled, with pre-test-post-test control group, follow-up) study. Both the mothers and fathers were included in the psychoeducation program for parents which was delivered in two sessions per week. The study was evaluated before the first session, after the second session and at the 6th month. Data were collected using the Personal Information Form and Caregiver Stress Scale (CSS). Mean, standard deviation, number and percentage, minimum, maximum, homogeneity tests and the chi-square test were used for data analysis.

DETAILED DESCRIPTION:
Psychoeducation given to the parents of the children with ADHD reduce parental stress, but these reduces are not proven for parents of the children with ADHD. The objective of this study was to determine the effect of psychoeducation on the stress levels of parents of children with Attention Deficit and Hyperactivity Disorder (ADHD). This was a randomised controlled study and applied the Consolidated Standards of Reporting Trials (CONSORT) statement. A total of 172 parents (experimental group: 86, control group: 86) participated in the study, which was planned as an experimental (randomized controlled, with pre-test-post-test control group, follow-up) study. Both the mothers and fathers were included in the psychoeducation program for parents which was delivered in two sessions per week. The study was evaluated before the first session, after the second session and at the 6th month. Data were collected using the Personal Information Form and Caregiver Stress Scale (CSS). Mean, standard deviation, number and percentage, minimum, maximum, homogeneity tests and the chi-square test were used for data analysis. The mean scores obtained from the scales before and after the training were compared with the paired-t test and student t test between the groups. There was no significant difference between the mean pre-test scores of the parents in the experimental and control groups on the whole CSS (p<0.005). Significant differences were found between the scores before and after the psychoeducation, and their six-month follow-up scores (p<0.001). There were significant differences between the pre- and post-test scores, pre-test scores and six-month follow-up scores, and post-test scores and six-month follow-up scores of the parents in the experimental group according to the in-group comparisons (p>0.05). It was determined that psychoeducation given to parents of children with ADHD reduced parental stress.

ELIGIBILITY:
Inclusion Criteria:

* having a child diagnosed with ADHD at least six months previously who was receiving standardized clinical follow-up and clinical treatment,
* being in the 18-65 age range,
* having no mental illness,
* agreeing to participate in the study

Exclusion Criteria:

* having a child without ADHD or having a child diagnosed with ADHD at least under six months previously who was receiving standardized clinical follow-up and clinical treatment,
* being younger 18 years and older 65 years,
* having a mental illness,
* agreeing not to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Caregiver Stress | 6 months
  The parents stress levels were evaluated with Caregiver Stress Scale. The data collected from experimental group before and after psychoeducation program and 6 months later. However, parents in control group had pretest and posttest at 6 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Gül Dikeç, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Gül Dikeç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided